CLINICAL TRIAL: NCT06948266
Title: Frequency and Clinical Features of Out-of-hospital Cardiac Arrest and Cardiopulmonary Resuscitation in 2023 in Poland - Retrospective Analysis.
Brief Title: The Study Aims to Investigate the Frequency and Clinical Characteristics of Out-of-hospital Cardiac Arrests (OHCA) Occurring in Poland in 2023. This Research Seeks to Provide a Comprehensive Analysis of OHCA Incidents Across the Country, Focusing on Their Prevalence and the Associated Clinical fe
Acronym: OHCA_PL
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Michal Szymanski, phd, Medical University of Gdansk
Other Study IDs: OHCA_PL
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Complications; Sudden Cardiac Arrest; Cardiac Diseases; Cardiac Arrest (CA)
Keywords: sudden cardiac death; poland; OHCA
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Diseases; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OHCA: OHCA in Oland in 2023.

SUMMARY:
1. Objective

   According to the 2021 European Resuscitation Council (ERC) Guidelines, sudden cardiac arrest is the third leading cause of death in Europe. Accurate and reliable data on the epidemiology of sudden cardiac arrest are essential for better understanding its causes and for analyzing treatment outcomes. Currently, comprehensive statistics on cardiac arrest in Poland are unavailable, resulting in limited knowledge about the scale of this medical issue. This study aims to examine the frequency and clinical characteristics of out-of-hospital cardiac arrests occurring nationwide in 2023.
2. Materials and Methods

   The analysis will include Emergency Medical Activity Cards from the year 2023. Data for the study will be obtained from the National Center for Monitoring Emergency Medical Services via the Department of Emergency Medical Services of the Polish Ministry of Health and from the Polish Medical Air Rescue. Data will be anonymized by data administrators before being provided to the research team.

   The analysis of the obtained results will be supplemented with publicly available data from the Central Statistical Office (GUS).

   The analyzed Emergency Medical Activity Cards will be evaluated according to the Utstein Out-of-Hospital Cardiac Arrest Registry template from 1991, with subsequent updates, the latest being in 2024, published under the title: "Cardiac arrest and cardiopulmonary resuscitation outcome reports: 2024 update of the Utstein Out-of-Hospital Cardiac Arrest Registry template - ILCOR Scientific Statement."
3. Study Population

   Adults who experienced out-of-hospital cardiac arrest in 2023.
4. Inclusion and Exclusion Criteria

   Exclusion Criteria:

   Age under 18 years.

   Inclusion Criteria:

   Emergency Medical Activity Cards containing at least one of the following criteria:

   In section IV DIAGNOSIS with ICD-10 codes: I46, R98, R96. In section III EXAMINATION, interview data indicating that bystanders initiated CPR.

   ResearchGate
   * 1 PMC
   * 1 In the SYMPTOMS table, marked as cardiac arrest. In the ECG table, marked rhythms: VF/VT, Asystole, PEA. In the PATIENT MANAGEMENT table, marked: MANUAL CHEST COMPRESSIONS, MECHANICAL CHEST COMPRESSIONS, DEFIBRILLATION.

   In the DEATH-WITHDRAWAL table, information on the reason for discontinuing resuscitation efforts.

   Only adult patients will be included in the study. Available demographic data will include patient age, gender, and the territorial area of the medical event, indicated by the location of the call and the voivodeship.
5. Estimated Study Group Size

   100,000 records.
6. Estimated Study Duration

The study is planned for a period of 6 months.

References:

European Resuscitation Council Guidelines 2021.

Gräsner JT, Bray JE, Nolan JP, et al. "Cardiac arrest and cardiopulmonary resuscitation outcome reports: 2024 update of the Utstein Out-of-Hospital Cardiac Arrest Registry template - ILCOR Scientific Statement."

DETAILED DESCRIPTION:
Frequency and Clinical Characteristics of Out-of-Hospital Cardiac Arrest in Poland in 2023

Background and Objective

Out-of-hospital cardiac arrest (OHCA) is a major public health concern and, according to the 2021 European Resuscitation Council guidelines, sudden cardiac arrest is the third leading cause of death in Europe cprguidelines.eu

. Despite its significance, Poland lacks a comprehensive national registry for OHCA, and complete nationwide data have not been available. This study is designed to fill that gap by determining the incidence of OHCA in Poland during 2023 and describing the clinical characteristics of these cases.

Methods

Study Design: This is a retrospective observational study analyzing all OHCA events that occurred in Poland in the year 2023. The study will use de-identified patient data drawn from official emergency medical service records. Data Sources: OHCA cases will be identified from the Emergency Medical Procedure Records (Karty Medycznych Czynności Ratunkowych, KMCR) for 2023. These records will be obtained through the National Emergency Medical Services Monitoring Center in collaboration with the Ministry of Health and the Polish Medical Air Rescue. All records will be anonymized by the data providers before being released to the research team to ensure patient confidentiality. In addition, publicly available demographic statistics from Statistics Poland (GUS) will be incorporated to provide context regarding population and regional distribution. Data Analysis: The collected data will be analyzed following the standardized Utstein-style template for reporting cardiac arrest, using the latest 2024 update for out-of-hospital cardiac arrest registries (as recommended by the International Liaison Committee on Resuscitation). This framework will ensure consistent definitions and allow benchmarking against international data. Key variables to be examined include the frequency (incidence) of OHCA, patient demographics (such as age and sex), circumstances of the arrest (e.g. location, whether it was witnessed, initial ECG rhythm), the interventions performed by bystanders and emergency medical services (such as CPR and defibrillation), and patient outcomes (including return of spontaneous circulation and survival to hospital admission). By adhering to the Utstein reporting guidelines, the study's findings will be comparable with other regional and international OHCA data, thereby enhancing their utility for epidemiological insight.

Significance

This study will provide the first comprehensive overview of OHCA occurrences across Poland for an entire year. The results are expected to furnish critical epidemiological data on how often cardiac arrests happen outside of hospitals and what clinical factors characterize these events. Such information is essential for public health authorities and medical professionals to understand current gaps in the chain of survival, to plan targeted interventions, and to improve resuscitation outcomes. Ultimately, the knowledge gained from this nationwide analysis can guide policy and training initiatives aimed at reducing mortality from sudden cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

Adults (≥18 years) who experienced an OHCA in 2023, identified through MEPCs containing at least one of the following indicators:

ICD-10 codes: I46, R98, R96 in the diagnosis section. Witness-reported initiation of CPR in the patient examination section. Indication of cardiac arrest in the symptoms table. Documented rhythms such as VF/VT, asystole, or PEA in the ECG table. Noted interventions like manual/mechanical chest compressions or defibrillation in the patient management table.

Reasons for cessation of resuscitation efforts in the death/discontinuation table.

Exclusion Criteria:

Individuals under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) who experienced an OHCA in 2023, identified through MEPCs
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
OHCA | 1 year
  Number of OHCA in Poland in 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Yes
Yes, individual participant data (IPD) that underlie the results reported in this study will be made available upon reasonable request. Interested researchers may contact the corresponding author via email to obtain access, contingent upon appropriate data use agreements and ethical approvals.
Supporting Information: Study Protocol, SAP
Time Frame: From 12.2025
Access Criteria: Who will have access:
  Access will be granted to researchers affiliated with academic institutions, hospitals, or other non-commercial research organizations, who demonstrate a legitimate scientific interest in the study topic. All requestors must have appropriate ethics approval for secondary data use if required by their institution or jurisdiction.